CLINICAL TRIAL: NCT06412445
Title: Self-Fixating Mesh Versus Mesh Fixation With Tissue Glue in Laparoscopic Transabdominal Inguinal Hernia Repair: A Comparative Study
Brief Title: Self-Fixating Mesh Versus Mesh Fixation With Tissue Glue in Laparoscopic Inguinal Hernia Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Adham Ashraf Maher Farid, General Surgery Assistant Lecturer, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mesh Fixation Methods in TAPP
Record Dates: First submitted 2024-04-03; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Inguinal Hernia
Keywords: TAPP; Self-Fixating Mesh; Mesh Fixation; Tissue Glue; Laparoscopic Transabdominal Inguinal Hernia Repair; Inguinal Hernia Repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetra-4-amidinophenoxypropane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with unilateral inguinal hernia undergoing TAPP repair and mesh fixation with tissue glue (Active Comparator): Patients aged from 18 to 60 years with unilateral direct or indirect inguinal hernia who will undergo laparoscopic TAPP inguinal hernia repair having there mesh fixated with tissue glue. Glubran 2® surgical glue is a medical device Class III CE marked for internal and external use. It is a synthetic biodegradable cyanoacrylate basis glue, modified by the addition of a monomer synthesized by the manufacturer GEM. It is ready for use. It has high adhesive and haemostatic properties and once it is polymerised it creates an efficient antiseptic barrier against the most diffused infective or pathogenic agents during the surgical intervention. It polymerizes quickly in contact with live tissue and wet environment creating a thin and elastic film having high tensile properties which guarantee strong adhesion to the tissues. This film naturally conforms with the tissues on which it is applied; it is not permeable to liquids and is not altered by blood or organic liquids
  Interventions: Procedure: Laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair applying tissue glue for mesh fixation
- Patients with unilateral inguinal hernia undergoing TAPP repair with self fixating mesh (Active Comparator): Patients aged from 18 to 60 years with unilateral direct or indirect inguinal hernia who will undergo laparoscopic TAPP inguinal hernia repair with self fixating mesh. Covidien ProGrip mesh is a self-gripping polyester mesh, 15x15 cm in size, it is equipped with resorbable microgrip technology which provides immediate fixation of the entire mesh surface for a secure repair and even distribution of tension for patient comfort. The resorbable polylactic acid (PLA) microgrips enable surgeons to position and place the mesh in under 60 seconds, without the use of additional fixation. Surgeons and patients can depend on a secure repair with the potential for greater patient comfort. According to the manufacturer, the time for degradation of the quickly absorbing layer is < 1 day and that for the layer with microgrips > 18 months
  Interventions: Procedure: Laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair using self-fixating mesh

INTERVENTIONS:
Procedure: Laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair applying tissue glue for mesh fixation — The operation will be performed using 3 trocars, with 10 mm trocar above the umbilicus and 5 mm and 12 mm trocars at the level of the umbilicus in the left and right midclavicular lines. Pneumoperitoneum will be established and a 30° optic will be used. After accessing the inguinal region, dissection of the parietal peritoneum will be performed in the direction from the anterior superior iliac spine up to the medial umbilical ligament. During dissection, gonadal vessels, vas deferens, Cooper's ligament and the posterior fascia of the rectus abdominis muscle will be visualized and prepared. Then, the prepared implant sized 15×15 cm will be introduced, spread out in the abdominal cavity and placed in the groin in order to cover the hernia opening by 2-3 cm in all directions. Fixation will be based on a mechanical effect involving applying tissue glue for mesh fixation. Reconstruction of the parietal peritoneum will be followed, with continuous absorbable sutures.
  Arms: Patients with unilateral inguinal hernia undergoing TAPP repair and mesh fixation with tissue glue
Procedure: Laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair using self-fixating mesh — The operation will be performed using 3 trocars, with 10 mm trocar above the umbilicus and 5 mm and 12 mm trocars at the level of the umbilicus in the left and right midclavicular lines. Pneumoperitoneum will be established and a 30° optic will be used. After accessing the inguinal region, dissection of the parietal peritoneum will be performed in the direction from the anterior superior iliac spine up to the medial umbilical ligament. During dissection, gonadal vessels, vas deferens, Cooper's ligament and the posterior fascia of the rectus abdominis muscle will be visualized and prepared. Then, the prepared implant sized 15×15 cm will be introduced, spread out in the abdominal cavity and placed in the groin in order to cover the hernia opening by 2-3 cm in all directions. Fixation will be based on a mechanical effect involving the adherence of grips to tissue using self-fixating mesh. Reconstruction of the parietal peritoneum will be followed, with continuous absorbable sutures.
  Other Names: TAPP procedure
  Arms: Patients with unilateral inguinal hernia undergoing TAPP repair with self fixating mesh

SUMMARY:
The main objective of this study is to compare between the safety and efficacy of self-fixating mesh versus mesh fixation with tissue glue in patients undergoing laparoscopic transabdominal inguinal hernia repair (TAPP). The criteria of comparison shall include operating time, post-operative pain and recurrence.

DETAILED DESCRIPTION:
Inguinal hernia is the most common abdominal wall hernia. It is defined as a peritoneal sac protrusion through a weak point within the groin area. It often contains abdominal contents and is traditionally treated with surgery. Repair of inguinal hernia is one of the most commonly performed surgical procedures worldwide. Males are more commonly affected by inguinal hernia than females. The male to female ratio is approximately 9 to 1.

Whether to perform an open or a laparoscopic approach for inguinal hernia repair has always been a controversial issue. However, recent improvement in laparoscopic techniques has made it the procedure of choice in the opinion of most surgeons. Laparoscopic approach includes two main techniques, namely the total extra-peritoneal approach (TEP) and the trans abdominal pre-peritoneal approach (TAPP). However, TAPP has gained more popularity owing to its relative simplicity and easier reproducibility. TAPP involves standard laparoscopic approach with access into the peritoneal cavity and placement of a mesh along the anterior abdominal wall, thereby, repairing the hernia posterior to the defect.

During the repair of an inguinal hernia, sutures or tacks are generally used to secure the prosthetic mesh in place. In TAPP repairs, the peritoneum is closed using sutures or tacks. These mesh fixation or peritoneal closure techniques may contribute to postoperative chronic pain presumably due to nerve irritation or entrapment. Intraoperative strategies to reduce pain entail the use of non-mechanical methods of mesh fixation other than tacking or suturing, which may be less traumatic to the local tissue and less likely to cause local nerve entrapment. These non-mechanical methods include self-fixating meshes or glue. Similarly, closing the peritoneum with sutures may be less traumatic than the use of tacks, thus resulting in less postoperative pain.

By far, guidelines of the European Association for Endoscopic Surgery (EAES) and the European Hernia Society (EHS) reported no general evidence based consensus on the ideal tool for mesh fixation. Therefore, the choice often depends on surgeons personal preference, market availability and cost/benefit ratio. Recent advances in the biotechnology of mesh and mesh fixation industry lead to the production of innovative self-fixating meshes and alternatively meshes that are fixed with variable types of biomaterials and glue. Eventually, such tack free meshes are intended to reduce the rate of complications that might be attributed to tack bearing meshes. However, studies to evaluate the different tools of tack free mesh fixation techniques are still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral direct or indirect inguinal hernia

Exclusion Criteria:

* Bilateral hernia.
* Femoral hernia.
* Inguinoscrotal hernia.
* Complicated inguinal hernias.
* Recurrent inguinal hernias.
* Morbid obesity.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | Follow up of all patients will be done post-operatively as outpatients after discharge on day 15, and after 3, 6 and 12 months
  clinical or radiological at any time point
Chronic pain | Follow up of all patients will be done post-operatively as outpatients after discharge on day 15, and after 3, 6 and 12 months
  pain persisting beyond three months postoperatively. Post-operative pain will be evaluated based on the numerical rating scale (NRS) 0-10, for pain self-reporting with reference to the patient's individual experience, where 0 indicates no pain, 1-3 mild pain, 4-6 moderate pain and 7-10 disabling severe pain

SECONDARY OUTCOMES:
Length of surgery | 1 to 3 hours
  in minutes
Immediate postoperative pain | 1 to 3 days
  Post-operative pain will be evaluated based on the numerical rating scale (NRS) 0-10, for pain self-reporting with reference to the patient's individual experience, where 0 indicates no pain, 1-3 mild pain, 4-6 moderate pain and 7-10 disabling severe pain
Vascular/visceral injury | 1 to 3 hours
  Any visualized or reported vascular or visceral injury during the operation
Haematoma/seroma development | 1 to 7 days
  Haematoma or seroma development in postoperative period (Clinical or radiological)
Length of hospital stay | 1 to 7 days
  in days
Urinary retention | 1 to 2 days
  in immediate postoperative period
Wound infection/mesh infection | 1 to 30 days
  at any time point
Recovery time to normal activity | 1 to 7 days
  in days

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No